CLINICAL TRIAL: NCT00005668
Title: A Multicenter, Prospective, Randomized, Double-Blind Clinical Trial Comparing Itraconazole Oral Solution in Cyclodextrin to Placebo in the Treatment of Aspergilloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: DMID MSG 37; DMID 96-199; NIH/09021
Record Dates: First submitted 2000-05-18; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Aspergillosis; Lung Diseases, Fungal
MeSH Terms: conditions — Aspergillosis; Lung Diseases, Fungal | interventions — Itraconazole

INTERVENTIONS:
Drug: Itraconazole oral solution

SUMMARY:
To compare the safety and effectiveness of itraconazole oral solution to placebo in the treatment of a pulmonary aspergilloma.

Aspergilloma is a "fungal ball" in the lungs caused by Aspergillus. The infection can spread from the lungs through the blood to other organs. Aspergilloma can be life-threatening; therefore, an effective treatment is needed.

DETAILED DESCRIPTION:
Patients are randomly selected to receive itraconazole oral solution by mouth or the inactive placebo (oral cyclodextrin solution) twice daily for 12 months.

ELIGIBILITY:
Inclusion Criteria:

You may be eligible for this study if you:

* Are 18 years of age or older.
* Have been diagnosed with aspergilloma within the last month.
* Have (or have a history of) at least one of the following:

  1. positive test for Aspergillus species.
  2. presence of antibodies to Aspergillus.
* Are willing to participate in the study for 2 full years.
* Are female and not pregnant.
* Are not breast-feeding.
* Agree to use barrier methods of birth control / contraception during the study and for 30 days after.

Exclusion Criteria:

You will not be eligible for this study if you:

* Have a history of allergy to triazole or imidazole drugs.
* Are unable to take oral medication.
* Are not expected to live for more than a month.
* Have had a lung biopsy indicating Aspergillus infection.
* Have had radiation therapy within the last 6 months.
* Require treatment with certain medications.
* Received amphotericin, amphotericin lipid formulation, fluconazole, or itraconazole in the two weeks prior to study entry.
* Received chemotherapy within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96
Dates: Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Ellen Bradley, Birmingham, Alabama, United States